CLINICAL TRIAL: NCT01242046
Title: The Effects of Caffeine on Female Genital Arousal
Brief Title: Effects of Caffeine on Women's Sexual Arousal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Key personnel were reassigned to different project
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Tierney Kyle Ahrold Lorenz, Researcher, University of Texas at Austin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2010-07-0070
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Sexual Behavior
Keywords: female sexual arousal
MeSH Terms: conditions — Sexual Behavior | interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Caffeine (Experimental): Participants will ingest a tablet with 400 mg caffeine
  Interventions: Dietary Supplement: Caffeine
- Placebo (Placebo Comparator): Participants will ingest an inert placebo tablet
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — 400 mg of caffeine in tablet form
  Arms: Caffeine
Dietary Supplement: Placebo — Inert tablet
  Arms: Placebo

SUMMARY:
The key research question in this study is whether or not caffeine facilitates genital sexual arousal in women in the presence of an external erotic stimulus. Caffeine's impact on the human sexual response cycle has yet to be studied in the field, so the goal is to determine if this substance will have any impact on genital arousal well as potentially identify the mechanisms underlying its ability to do so. Considering that this will be a single blind study, a key goal of the project is to determine how participant expectations regarding what they ingest will impact their subjective sexual arousal. At present, we hypothesize that, as caffeine's stimulant properties increase a human's heart rate and blood pressure, caffeine intake will facilitate genital arousal.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 or older
* Heterosexual
* Experiencing regular menstrual cycles (not more than 1 missed menstrual period in the past 6 months).
* Currently involved in a stable, sexually active relationship.
* Fluent in the English language.

Exclusion Criteria:

* Self-report of sexual aversion or distress; or of distress related to a history of unwanted or coercive sexual contact.
* Perimenopausal or menopausal status, or >1 missed menstrual period in the previous 6 months; or currently pregnant, breastfeeding, or having breastfed within the past 3 months; or clinically significant untreated renal or endocrine disease.
* History of HIV infection or active, untreated pelvic, vaginal, or urinary tract infection including sexually transmitted diseases such as chlamydia, genital herpes, gonorrhea, or syphilis.
* Previous major pelvic surgery that may have caused nerve damage, including hysterectomy, vulvectomy, circumcision, colostomy, cystostomy, or serious bladder, rectal, or abdominal surgery; or neurological impairment due to diabetes, stroke, pelvic nerve damage secondary to trauma, cancer treatments, myasthenia gravis, multiple sclerosis or spinal cord damage.
* Self-report of an untreated psychosis (e.g., bipolar disorder or schizophrenia).
* Women who do not use caffeine products regularly (i.e., on a daily basis).
* Women receiving any of the following medications will be excluded from the study, as they have been shown to alter sexual function or arousal response: Dehydroepiandrosterone (DHEA), testosterone and other androgens, estrogens (except oral contraceptives), progesterone, tamoxifen, raloxifene, and other selective estrogen receptor modulators (SERMs), Beta blockers or other drugs that affect the autonomic nervous system and/or cardiovascular system, any approved or experimental medications or treatments used to enhance the sexual response (e.g., sildenafil), and antidepressants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Sexual arousal | 15 minutes post administration of drug or placebo
  Vaginal pulse amplitude, as measured by a vaginal photoplethysmograph

CONTACTS AND LOCATIONS:
Overall Officials: Corey A Pallatto, B.A., Principal Investigator — University of Texas at Austin
Locations (1):
- University of Texas at Austin, Austin, Texas, United States

REFERENCES:
- See also: Laboratory website — http://www.mestonlab.com